CLINICAL TRIAL: NCT03067467
Title: Investigating Metabolic Characteristics of Intracranial Malignancy in Vivo Using Hyperpolarized Carbon-13 Magnetic Resonance Spectroscopic Imaging (MRSI)
Brief Title: Metabolic Characteristics of Brain Tumors Using Hyperpolarized Carbon-13 Magnetic Resonance Spectroscopic Imaging (MRSI)
Acronym: HPCIM
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jae Mo Park, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 012017-070
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Brain Tumor Adult
MeSH Terms: interventions — Gadolinium; gadobutrol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Brain Tumor Patients: Brain Tumor patients will receive a bolus of Hyperpolarized 13C-pyruvate during MRSI.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate; Drug: Gadolinium

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Hyperpolarized 13C-pyruvate IV bolus followed by brain MRSI.
  Other Names: HP [1-13C]pyruvate
Drug: Gadolinium — Brain MRI performed with and without gadolinium-based contrast.
  Other Names: Gadavist

SUMMARY:
This is a non-randomized, purely observational, feasibility study to detect metabolic changes in patients with brain malignancy using a novel hyperpolarized [1-13C]pyruvate MRSI.

DETAILED DESCRIPTION:
The aim of this pilot study is to test the hypothesis that patients with brain malignancy present altered [1-13C]lactate and 13C-bicarbonate production from infused hyperpolarized [1-13C]pyruvate in tumor as compared to in normal-appearing brain regions. To achieve this aim investigators will assess metabolic phenotype in cancer patients with brain tumors (n = 20). Total target enrollment will be set at 25 subjects to account for attrition and screening failures.

During each imaging session, following localization of the tumor in brain, tissue characteristics and morphological changes will be evaluated with 1H MRI. Then, cerebral metabolism will be assessed utilizing 13C MRSI after an intravenous injection with hyperpolarized [1-13C]pyruvate. Finally, contrast-enhanced 1H MRI will be acquired. The study agent, hyperpolarized [1-13C]pyruvate, will be administered under a Food and Drug Administration (FDA) Investigational New Drug (IND), which was approved on 1/3/2017 (IND# 133229).

Preliminary data in human are essential to secure larger scale funding required for clinical studies. The investigators believe the ability to measure such metabolic shifts in vivo could have major significance in assessing the efficacy of multiple anti-tumor therapies currently under development that target reversing the Warburg effect as a means of controlling tumor growth. Brain tumor applications at the Advanced Imaging Research Center, Harold C. Simmons Comprehensive Cancer Center and the Neuro-Oncology Program of the Development of Neurological Surgery at the UT Southwestern Medical Center offer today a unique opportunity to lead globally the translational scientific efforts in this field.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of brain tumors by imaging which demonstrates all kinds of brain malignancy, including glioma, meningioma, and brain metastases prior to any chemotherapy or radiation treatment.
* 18-70 years of age
* Ability to understand and the willingness to sign a written informed consent.
* All races and ethnicities will be included; subjects must be able to read and speak the English language. Once the protocol is established, Spanish-speaking participants will be included.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Subjects who are receiving any other investigational agents.
* Previous or current treatment by radiation or chemotherapy.
* Concurrent illness including, but not limited to, ongoing or active infection, uncontrolled chronic diseases such as hypertension, lung disease, liver disease, kidney disease, diabetes, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects who have a history of alcohol abuse or illicit drug use.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* Subjects who have contraindication to contrast enhanced MRI examination

Contraindications to MRI examination include:

* Medically unstable

  * Heart failure
  * Severe LVOT outflow obstruction
  * Unstable angina
  * Child bearing
  * Lactating
* Any contraindication per MRI Screening Form including

  * Implants contraindicated at 3T, pacemakers
  * Implantable Cardioverter Defibrillator (ICD)
  * Claustrophobia
* Since each subject may be receiving a gadolinium-based contrast agent intravenously:

  * eGFR ≤ 30 mL/min/1.73m2
  * Sickle cell disease
  * Hemolytic anemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 Brain Tumor Patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
13C-pyruvate Metabolic Product Ratio | Screening (Baseline) and 1 day of Study Visit
  Measurement of the ratio of metabolic products, [1-13C]lactate and 13C-bicarbonate, from hyperpolarized [1-13C]pyruvate will be used as an index of metabolic balance between glycolytic pathway and mitochondrial oxidative phosphorylation.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Mo Park, PhD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No